CLINICAL TRIAL: NCT06692530
Title: Paranoid Behaviour & Threat Evaluation in Asylumseekers Diagnosed With a Psychotic Disorder and Experiencing Paranoid Delusions: A Phenomenological Qualitative Virtual Reality Study
Brief Title: Asylumseekers Experiencing Paranoid Delusions: A Virtual Reality Study
Acronym: COA-VR
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: NL84630.042.23
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-11

CONDITIONS: Schizophrenia Disorders; Paranoid Delusions
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Rationale: Ethnic minorities and asylumseekers have a two- to three-times increased risk of psychosis compared to people from their host country. Among patients experiencing psychosis, paranoid delusions are a common symptom. Diagnostic assessments are challenging in this group because of language differences and sociocultural differences in interpersonal social behavior and communication. To fill this gap this research will make use of Virtual Reality (VR) to assess thoughts, behaviours and emotions in real-time. VR has a high ecological validity and its partial non-verbal nature has a clear potential in terms of a transcultural application among asylumseekers.

Objective: The main objective of this study is to discover how asylumseekers with a psychotic disorder who are experiencing paranoid delusions behave and evaluate threat in a virtual environment.

Secondary objectives: To assess the suitability and applicability of using VR within the specific population of asylumseekers with a psychotic disorder and paranoid delusions.

Study design: The study uses a mixed-methods design, combining qualitative phenomenological data and descriptive quantitative data.

Study population: Adult psychiatric patients that are seeking asylum in the Netherlands with a DSM-5 classification of a psychotic disorder and paranoid delusion (as measured by the PANSS) will be included. Furthermore, patients must receive mental health care from CTP Veldzicht, either in one of the wards (closed or open) or through ambulatory care.

Intervention: The patients will be immersed in a VR-environment using a head mounted display. Four different VR-scenarios are used, each taking up three to four minutes. Using simple movement instructions, patients are asked to walk around and observe their environment.

Main study parameters/endpoints: Phenomenological semi-structured interview. The interview measures the experience of participants in a qualitative matter. Audio recordings of the semi-structured interviews will be transcribed. These transcriptions containing rich qualitative data are the main study parameter. Additional descriptive qualitative data (demographic & symptom specific) will be gathered through questionnaires to provide quantitative insight in the sample-population (questionnaires used: PANSS, SSPS, SBQ, and VAS). Subsequently, psychiatrists working in the field of transcultural psychiatry will be interviewed about the paranoid behaviour of participants based on video and audio recordings of the VR-session.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Some participants might experience simulator sickness symptoms. No major adverse events are expected or have been documented in previous VR studies of our research group using the same VR hardware and software. The assessment will take approximately 90 minutes in total. No benefits are expected. An empathic and transparent approach, a clear consent procedure, close monitoring of participants' moods and consistently adverting an opt-out will be used.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Receiving treatment from CTP Veldzicht
* Seeking asylum in the Netherlands, registered with Centraal Opvang Asielzoekers (COA)
* Classification (primary or subsidiary classification) of a disorder categorized within the 'schizophreniaspectrum- and other psychotic disorders' (DSM-V)
* Diagnosed with the symptom of paranoid delusion, defined as a PANSS score on the delusion item (P6) >2

Exclusion Criteria:

* Unable to provide informed consent
* Acutely psychotic, which means overwhelmed by psychotic symptoms, agitated, not able to participate in an interview, as judged by a therapist or socio-therapist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be recruited from departments within the Centre for Transcultural Psychiatry Veldzicht. These departments consist of three closed-wards, one open ward, and a department that provides ambulatory-care in asylumseeker centres in the northeast of the Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Phenomenological qualitative interview Data | One data collection moment per participant which takes 2.5 hours.
  The interview measures the experience of participants in a qualitative matter. Audio recordings of the semi-structured interviews will be transcribed. These transcriptions containing rich qualitative data are the main study parameter.

CONTACTS AND LOCATIONS:
Locations (1):
- CTP Veldzicht, Balkbrug, Overijssel, Netherlands